CLINICAL TRIAL: NCT00795483
Title: Efficacy and Security of Annual and Biennial Zoledronic Acid for Osteoporosis Treatment in an HIV-infected Patients' Cohort
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Dra. EUGENIA NEGREDO PUIGMAL, Eugenia Negredo, Germans Trias i Pujol Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIH-ZOL
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2012-08

CONDITIONS: HIV Infections
Keywords: Osteoporosis; HIV infection; Bisphosphonates; Zoledronic acid
MeSH Terms: conditions — HIV Infections; Osteoporosis | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1-ANNUAL (Experimental): 1. Zoledronic acid + Lifestyle modifications (experimental)
  Interventions: Drug: Zoledronic acid; Behavioral: Lifestyle modifications
- 2-CONTROL (Other): 2. Lifestyle modifications (control)
  Interventions: Behavioral: Lifestyle modifications
- 3-BIENNIAL (Experimental): 3. Zoledronic acid + Lifestyle modifications (experimental)
  Interventions: Behavioral: Lifestyle modifications; Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid — Zoledronic Acid 5mg/year
  Arms: 1-ANNUAL
Behavioral: Lifestyle modifications — Lifestyle modifications
Drug: Zoledronic acid — Zoledronic acid (5mg/2years)
  Arms: 3-BIENNIAL

SUMMARY:
The purpose of this project is to determine the incidence of osteoporosis in the investigators' population of HIV-infected patients and to assess the efficacy and security of zoledronic acid, whose efficacy in post-menopausal women with high fracture risk treatment and in Paget's disease treatment has already been demonstrated.

DETAILED DESCRIPTION:
The lower bone mineral density that has been described in patients with HIV-infection has not meant an increase of long term complications. Nevertheless, it could involve an increase if the associated co-morbidity in the future, taking in care that in general population osteoporosis increases 4 times the pathologic fracture risk. That is why it is necessary to know the real prevalence of osteoporosis in this population of patients so the real dimensions of the problems can be defined.

This project wills to determine the incidence of osteoporosis in our population of HIV-infected patients and to assess the efficacy and security of zoledronic acid. If the annual use of endovenous zoledronic acid obtains equivalent results to those obtained with oral and weekly alendronate in other studies with the same population, its use would be justified because of its posology benefits. The annual administration can improve compliance in patients who are receiving a big quantity of drugs, as HIV-infected patients do, and who probably have to be treated for life. Moreover, its elimination is renal so there is absence of interactions with antiretroviral drugs what makes of zoledronic acid a very promising alternative. Finally, there is no risk of digestive intolerance because of its parenteral administration and it has a better posology than oral bisphosphonates.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older.
2. Documented HIV-1 infection, with or without antiretroviral treatment.
3. Presence of WHO osteoporosis criteria, defined as t-score under -2.5 in lumbar, hip and/or trochanter (DEXA in the last 6 months is needed).
4. Willing to follow the study protocol.
5. Informed Consent signature.

Exclusion Criteria:

1. In women, pregnancy or breastfeeding.
2. Other possible causes of secondary osteoporosis.
3. Creatinine over 2.3 mg/mL.
4. Glomerular filter less than 50 mL/min (estimated through MDRD).
5. Treatment for Osteoporosis in the last 4 months.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Increase in lumbar (L2-4) and femoral (trochanter, femur neck, total femur and hip) t-score bone mineral density | Evolution from baseline to week 48
Increase in lumbar (L2-4) and femoral (trochanter, femur neck, total femur and hip) t-score bone mineral density | Evolution from baseline to week 96

SECONDARY OUTCOMES:
Adverse events | From baseline to week 96
Lab tests | Evolution from baseline to week 96
Related clinical events (bone fractures) | From baseline to week 96
Osteoblastic/Osteoclastic activity, bone formation/reabsorption. | Evolution from baseline to week 48
Osteoblastic/Osteoclastic activity, bone formation/reabsorption. | Evolution from baseline to week 96

CONTACTS AND LOCATIONS:
Overall Officials: Negredo Eugenia, MD,PhD, Principal Investigator — LLuita contra la SIDA Foundation
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain